CLINICAL TRIAL: NCT01430988
Title: An Observational Clinical Study of the BrainScope® Ahead™ M-100 Hand Held Electroencephalogram in Emergency Department Patients With Head Injury (B-AHEAD UK Trial)
Brief Title: Observational Study of the BrainScope® Ahead™ M-100 in UK Emergency Department Patients With Head Injury
Status: Terminated | Type: Observational
Why Stopped: The trial was terminated prematurely following a suspected data processing concern in the study device. The concern did not pose a patient safety issue.
Sponsor: BrainScope Company, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ahead™ M-100 B-AHEAD UK
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Brain Injuries; Craniocerebral Trauma
Keywords: Head Injuries; Head Trauma; TBI (Traumatic Brain Injury); Emergency Department; Accident & Emergency
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Brain Injuries, Traumatic; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Head Injured Group: Subjects who are suspected of a traumatically induced structural brain injury and/or clinical manifestations of functional brain injury, as a result of insult to the head from an external force, e.g., the head being struck by an object, the head striking an object, the head being exposed to forces generated from a blast or explosion, and/or the brain undergoing an acceleration/deceleration movement without direct external trauma to the head will be recruited from patients who enter the Emergency Department at hospitals that are participating as clinical sites for this study
- Normal Control Group: A normal control group will be recruited for comparison and will consist of Emergency Department patients who have sustained an injury but do not exhibit any trauma above the clavicle and no history of Road Traffic Accident requiring an ED visit or TBI within the past one (1) year, and no primary complaint of syncope.
- Head Injured Control Group: A 'head injured' control group will be recruited and will consist of Emergency Department patients who are suspected or who have sustained a head injury but do not report or manifest symptoms, e.g. facial lacerations and/or whiplash.

SUMMARY:
The purpose of the current study is proposed to prospectively assess how accurately the BrainScope® Ahead™ M-100 can distinguish risk categories for acute head injury.

DETAILED DESCRIPTION:
One million patients attend Emergency Departments (ED) with head injuries each year in the United Kingdom (UK) and Ireland. 150,000 of these patients will need hospital admission and one study estimates an incidence of 45-48% moderate or severe disability in those surviving admission. Although the incidence of head injury is high, the incidence of death from head injury is low. Therefore ED's are required to see a large number of patients with a minor/mild head injury, and identify the very small number of these that will go on to have serious complications. The challenge to the emergency medicine clinician is identifying which patients with a head injury have an important brain injury that requires further attention and which patients can be safely sent home. The standard for determining an important brain injury is the result on the Computerised Tomography (CT) scan of the head. CT scanning is nonportable and exposes individuals to high radiation levels.

The study medical device is a portable, point of care, noninvasive and non radiation-emitting medical device designed to assist clinicians in early identification, staging, and optimisation of treatment for patients who are head injured.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 to 80 (the entire age range), who are admitted to the Emergency Department (ED), who are suspected of a traumatically induced structural brain injury and/or clinical manifestations of functional brain injury, as a result of insult to the head from an external force, e.g., the head being struck by an object, the head striking an object, the head being exposed to forces generated from a blast or explosion, and/or the brain undergoing an acceleration/deceleration movement without direct external trauma to the head with a Glasgow Coma Scale of >8. The acute, suspected traumatically induced structural brain injury and/or clinical manifestations of functional brain injury will have occurred within the past 24 hours upon admission to the ED.
* The 'head injured' control group will be males and females ages 18 to 80 (the entire age range), who are admitted to the ED and are suspected or who have sustained a head injury but do not report or manifest symptoms, e.g. facial lacerations and/or whiplash.
* The ED normal control group will be males and females ages 18 to 80 (the entire age range), who are admitted to the ED for presenting complaints that do not involve the head or neck (no trauma above the clavicles) and no history of Road Traffic Accident requiring an ED visit or TBI within the last one (1) year and no primary complaint of syncope.

Exclusion Criteria:

* Subjects will be excluded who have forehead, scalp, or skull abnormalities or other conditions that would prevent correct application of the electrode headset on the skin. In addition, subjects with dementia, Parkinson's Disease, multiple sclerosis, seizure disorder, brain tumours, history of brain surgery, psychiatric disorder for which there is a prescribed psychiatric medication taken on a daily basis, substance dependence, history of TIA or stroke within the last year, currently receiving dialysis or in end-stage renal disease, active fever defined as greater than 100 degrees F or 37.7 degrees C, current condition is listed as "critical", subject is suffering from an open head injury, subject requires advanced airway management (i.e. mechanical ventilation), currently receiving procedural sedation medications (e.g. benzodiazepine, anaesthetic, NMDA receptor antagonist, or opioid agonist), subjects below the age of 18 years, pregnant women, and prisoners will not be eligible for study. ED normal control subjects will be excluded if there is a suspected neck injury or trauma above the clavicles, a primary complaint of generalized weakness, or a primary complaint of headache or migraine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the Emergency Department or Accident & Emergency within the selected hospitals participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Structural Injury Assessment | Within 24 hours of head injury
  There are four co-primary endpoints in this study: two sets of sensitivity and specificity to divide the data into three classes.
  Using a BrainScope classification algorithm, the Ahead M100 will identify subjects showing sensitivities among 3 classes: Green-normal, nonhead injured controls,Yellow-head injured subjects who do not exhibit brain electrical activity that is consistent with a structural brain injury observable on CT or for whom CT was not deemed necessary,Red-head injured subjects who exhibit brain electrical activity consistent with a structural brain injury observable by CT.

SECONDARY OUTCOMES:
Functional Injury Assessment | Within 24 hours of head injury
  There are two co-secondary endpoints for the secondary objective, the sensitivity and specificity to split Yellow from the primary endpoint into two sub groups depending on degree of brain functional impairment observable by an evaluation of the clinical findings on a clinical charter used as the assessment of truth.

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Pearse, MD, Principal Investigator — Royal London Hospital, Barts and The London School of Medicine and Dentistry
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, Cambridge
  - Royal London Hospital, Whitechapel, London
  - Salford Royal Hospital, Salford, Manchester

REFERENCES:
- [Background] Naunheim RS, Treaster M, English J, Casner T. Automated electroencephalogram identifies abnormalities in the ED. Am J Emerg Med. 2011 Oct;29(8):845-8. doi: 10.1016/j.ajem.2010.03.010. Epub 2010 May 1. PMID 20825903
- [Background] Naunheim RS, Treaster M, English J, Casner T, Chabot R. Use of brain electrical activity to quantify traumatic brain injury in the emergency department. Brain Inj. 2010;24(11):1324-9. doi: 10.3109/02699052.2010.506862. PMID 20722504
- [Background] Naunheim RS, Casner T. Novel method for detecting brain abnormality in a patient with epidural hematoma: a case report. Am J Emerg Med. 2010 Mar;28(3):386.e1-2. doi: 10.1016/j.ajem.2009.05.008. PMID 20223405
- [Background] McCrea M, Prichep L, Powell MR, Chabot R, Barr WB. Acute effects and recovery after sport-related concussion: a neurocognitive and quantitative brain electrical activity study. J Head Trauma Rehabil. 2010 Jul-Aug;25(4):283-92. doi: 10.1097/HTR.0b013e3181e67923. PMID 20611046